CLINICAL TRIAL: NCT03950570
Title: A Phase 1/2, Open Label, Dose-Escalation and Expansion Study of Oral ORIN1001 with and Without Chemotherapy in the Treatment of Subjects with Solid Tumors
Brief Title: ORIN1001 in Patients with Advanced Solid Tumors and Relapsed Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orinove, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORIN1001-001
Record Dates: First submitted 2019-04-23; First posted 2019-05-15 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor; Metastatic Breast Cancer
Keywords: Solid tumors, Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase 1: Dose escalation as a single agent (all tumor types); Dose escalation in combination with Abraxane (Breast Cancer);
  Phase 2: Dose expansion as a single agent or in combination with Abraxane (breast cancer)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1a: Dose Escalation with ORIN1001 (Experimental): In patients with advanced solid tumors or metastatic breast cancer: Treatment with a single oral agent, ORIN1001.
  Interventions: Drug: ORIN1001
- Experimental Phase 1b: Dose escalation - ORIN1001 in combination with Abraxane dose (Experimental): In patients with Relapsed, refractory metastatic breast cancer: Treatment with a combination of ORIN1001 and Abraxane.
  Interventions: Drug: Abraxane; Drug: ORIN1001

INTERVENTIONS:
Drug: Abraxane — In patients with relapsed. metastatic breast cancer, ORIN1001 will be administered in combination with Abraxane administered by intravenous infusion.
  Arms: Experimental Phase 1b: Dose escalation - ORIN1001 in combination with Abraxane dose
Drug: ORIN1001 — ORIN1001 will be administered as a table as a monotherapy in the dose escalation phase in patients with advanced solid tumors or in combination with Abraxane in patients with relapse, refractory breast cancer

SUMMARY:
This study evaluates the anti-tumor effects of ORIN 1001 in patients with advanced solid tumors or relapsed refractory metastatic breast cancer (patients with progressive disease after receiving at least two lines of therapy in the advanced setting).

DETAILED DESCRIPTION:
This is a first in human, Phase 1/2, open label, dose escalation and dose expansion study that consists of two stages:

Phase 1: A dose escalation stage to determine the MTD/RP2D of ORIN1001 when given as a single agent in up to 30 subjects with advanced solid tumors. In addition, a dose escalation stage to determine the MTD/RP2D of daily ORIN1001 in combination with Abraxane given intravenously in up to 18 subjects with relapsed refractory metastatic breast cancer (TNBC or ER+ HER2-).

Phase 2: An expansion stage of ORIN1001 alone (Cohort A: TNBC) and in combination with Abraxane (Cohort B: Myc+; Cohort C: ER+ HER2-, and Cohort D: TNBC) to estimate efficacy in up to 120 subjects with relapsed refractory metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

For dose escalation with ORIN1001 alone:

-Male or female with advanced solid tumors for which no effective standard of care treatments are available

For dose escalation with ORIN1001 in combination with Abraxane:

-Males or females with relapsed refractory metastatic breast cancer (TNBC or ER+, HER2-) must have progressed through at least 2 lines of therapy and for whom there are no available therapies that confer a clinical benefit

For dose expansion:

a. Males or females with relapsed refractory metastatic breast cancer including:

1. TNBC (i.e. estrogen receptor (ER)-, progesterone receptor-, and human epidermal growth factor receptor 2 [HER2]-)
2. ER+ HER2- breast cancer

Inclusion Criteria for Dose Escalation and Dose Expansion

1. Adults aged ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
3. Life expectancy of 3-4 months
4. Have at least one measurable lesion per RECIST 1.1
5. Have adequate organ function, including all of the following:

   1. Adequate bone marrow reserve as defined by: ANC≥1.0 x 10 9/L; platelet count ≥75 x 10 9/L; hemoglobin ≥9 g/dL
   2. Hepatic: total bilirubin ≤2 x ULN, transaminases (AST/SGOT and/or ALT/SGPT) ≤ 3X ULN;alkaline phosphatase ≤ 5 x ULN
   3. Renal: 24-hour creatinine clearance ≥ 30 mL/min calculated
6. Adequate tissue sample from either archival tumor tissue or fresh biopsy of tumor at the screening for tumor genotyping.
7. Male subjects must be surgically sterile or must agree to use physician approved contraception for 7 days prior to the first study drug administration to 30 days after the last dose of study treatment.
8. Women of childbearing potential must have negative serum pregnancy test within 14 days prior the first administration of study drug and agree to use physician-approved contraception from 30 days prior to the first study drug administration to 30 days following the last study drug administration.
9. Ability to understand and willingness to sign an informed consent prior to any study specific procedures.
10. Resolution of all toxicities (except alopecia) from prior therapy to ≤ Grade 1 (CTCAE v5)

Exclusion Criteria:

1. Does not meet inclusion criteria
2. Received any of the following within the specified time frame prior to the first administration of study drug:

   i. Excluding those with a history of coagulopathy ii. Excluding those who require concurrent use of anti-coagulants or anti-platelet medication, with exception of aspirin doses ≤ 81 mg/day, prophylaxis subcutaneous (SC) heparin or SC low-molecular weight heparin for deep vein thrombosis (DVT) prophylaxis or heparin flushes to maintain IV catherer patency iii. Excluding subjects that have Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastin time (aPTT) >1.5 x ULN b.Prior chemotherapy or other systemic anticancer therapy within 3 weeks or 5 times the plasma half-life of the drug, whichever is shorter; c.Prior radiotherapy within 2 weeks; d.Major surgery within 2 weeks; e.Prior treatment with investigational drugs within 4 weeks; f. Myocardial infarction, uncontrolled angina,severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, within 6 months prior to the fist dose of study drug
3. Greater than Class II heart failure using New York Heart Association (NYHA) criteria
4. The subject has uncontrolled human immunodeficiency virus (HIV) infection or active hepatitis B or C infection or other known active and/or uncontrolled infection
5. Active autoimmune disease that is not appropriately controlled with treatment
6. Active malignancy with the exception of:

   1. adequately treated basal cell carcinoma, squamous cell carcinoma, or in situ cervical cancer
   2. adequately treated stage I cancer from which the subject is currently in remission, or
   3. any other cancer from which the subject has been disease-free for ≥3 years;
7. Any serious uncontrolled medical or psychological disorder that would impair the ability to receive protocol therapy
8. Any condition which places the subject at unacceptable risk or confounds the ability of the investigator to interpret study data
9. The subject is pregnant or lactating woman. Any woman who becomes pregnant during the study will be withdrawn from the study.
10. Known active uncontrolled or symptomatic brain metastases. Patients with a history of such metastases that have been treated and are stable ≥28 days may be enrolled. Patients with no steroid use for at least 2 weeks prior to the time of enrollment are permitted.
11. Failed to respond to the most recent dose of Abraxane and must have been received at least 12 months prior to starting treatment.(combination arm only)
12. Greater than Grade 1 neuropathy (combination arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
To determine the safety of MTD/RP2D of single-agent daily ORIN1001 when administered orally in subjects with advanced solid tumors: NCI CTCAEv5 Common Toxicity Criteria | From first dose up to 21 days after last dose
  To determine the safety of the maximal tolerated dose/ recommended Phase 2 dose (MTD/RP2D). Incidence of the safety population will consist of all subjects who received a dose of study drug. Treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. Adverse events will be evaluated and recorded according to NCI CTCAEv5 Common Toxicity Criteria and will use medical terminology based on the Medical Dictionary for Regulatory Activities Terminology (MedDRA).
To determine the safety MTD/RP2D of daily ORIN1001 when administered orally in combination with paclitaxel given intravenously at 175 mg/m2 once every three weeks in subjects with relapsed refractory metastatic breast cancer | From first dose up to 21 days after last dose
  Incidence of the safety population will consist of all subjects who received a dose of study drug. Treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. Adverse events will be evaluated and recorded according to NCI CTCAEv5 Common Toxicity Criteria and will use medical terminology based on the Medical Dictionary for Regulatory Activities Terminology (MedDRA).
To evaluate the safety and tolerability of single-agent daily ORIN1001 when administered orally in the dose escalation and expansion stages of the study: NCI CTCAEv5 Common Toxicity Criteria | From first dose up to 21 days after last dose
  Incidence of the safety population will consist of all subjects who received a dose of study drug. Treatment-related AE is any untoward medical occurrence attributed to study drug in a participant who received study drug. Adverse events will be evaluated and recorded according to NCI CTCAEv5 Common Toxicity Criteria and will use medical terminology based on the Medical Dictionary for Regulatory Activities Terminology (MedDRA).
To evaluate the safety and tolerability of daily ORIN1001 when administered orally in combination with Abraxane given intravenously at 100 mg/m2 once weekly for 3 weeks in the dose escalation and expansion stages of the study | From first dose up to 28 days after last dose
  Incidence of number of participants with clinically significant change in vital signs. Vital signs include body weight, body temperature, resting blood pressure, pulse and respiratory rate.

SECONDARY OUTCOMES:
To evaluate the peak concentrations (Cmax) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent peak concentrations (Cmax) of ORIN1001 by direct inspection of the plasma concentration-time curves of ORIN1001 following single and repeat oral doses of ORIN 1001 as a single agent and in combination with Abraxane.
To evaluate the time to peak concentrations (Tmax) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent time to peak concentrations (Tmax) of ORIN1001 by direct inspection of the plasma concentration-time curves of ORIN1001 following single and repeat oral doses of ORIN 1001 as a single agent and in combination with Abraxane.
To evaluate the area under the plasma concentration versus time curve (AUC) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent area under the plasma concentration versus time curve (AUC) for ORIN1001 following single doses of ORIN 1001 as a single agent and in combination with Abraxane.
To evaluate the last time point with a quantifiable concentration (AUClast) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent plasma levels of ORIN1001 from the time of dosing to the last time point with a quantifiable concentration (AUClast) of ORIN1001 following single doses of ORIN 1001 as a single agent and in combination with Abraxane.
To evaluate the plasma concentration end of a dosing interval (Ctau) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent plasma concentrations (Cmax) of ORIN1001 as single agent or in combination with Abraxane at the end of a dosing interval (Ctau), where tau is 24 hours for once daily dosing.
To evaluate the average plasma concentration (Cav) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the average plasma concentration (Cav) of ORIN1001 as single agent or in combination with Abraxane during the dosing interval.
To evaluate the minimum plasma concentrations (Cmin) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the the minimum plasma concentrations (Cmin) reached by ORIN1001 as single agent or in combination with Abraxane prior to administration of a second dose.
To evaluate the elimination constant (λz) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent plasma elimination constant (λz) for ORIN1001 as a single agent or in combination with Abraxane.
To evaluate the terminal half-life (T1/2) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent terminal plasma half-life of ORIN1001 (T1/2) as a single agent or in combination with Abraxane.
To evaluate the plasma clearance (CL/f) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the dose-dependent apparent total plasma clearance (CL/f) of ORIN1001 after oral administration as a single agent or in combination with Abraxane.
To evaluate the volume of distribution (Vz/f) of ORIN1001 after oral administration as a single agent and in combination with Abraxane. | 2 months
  Determine the apparent volume of distribution (Vz/f) during terminal phase after oral administration of ORIN1001 as a single agent or in combination with Abraxane.

OTHER OUTCOMES:
To quantify the objective response rate (ORR) of ORIN1001 alone and in combination with Abraxane | Baseline up to approximately 2 years
  To quantify the proportion of patients with an objective tumor response as defined by RECIST 1.1 response criteria (SD, PR, CR).
To quantify the difference in the objective response rate (ORR) in relapsed refractory metastatic breast cancer showing potentially response-predictive aberrations of MYC and other genes under ORIN1001 alone or in combination with Abraxane | Baseline up to approximately 2 years
  To quantify the proportion of patients with an objective tumor response as defined by RECIST 1.1 response criteria (SD, PR, CR).
To measure the response duration in patients receiving ORIN1001 alone and in combination with Abraxane. | Baseline up to approximately 2 years
  To measure the duration of response from the time point of first established response (SD, PR, CR) until the time of documented tumor progression.
To quantify the difference in the duration of response in relapsed refractory metastatic breast cancer showing potentially response-predictive aberrations of MYC and other genes under ORIN1001 alone or in combination with Abraxane | Baseline up to approximately 2 years
  To measure the duration of response from the time point of first established response (SD, PR, CR) until the time of documented tumor progression.
To measure the time to response in patients receiving ORIN1001 alone and in combination with Abraxane. | Baseline up to approximately 2 years
  To measure the time from cycle 1 day 1 dose to the time of first documentation of tumor response (SD, PR, CR).
To quantify the difference in the time to response in relapsed refractory metastatic breast cancer showing potentially response-predictive aberrations of MYC and other genes under ORIN1001 alone or in combination with Abraxane. | Baseline up to approximately 2 years
  To measure the time from cycle 1 day 1 dose to the time of first documentation of tumor response (SD, PR, CR).
To measure the duration of progression free survival (PFS) in patients receiving ORIN1001 alone and in combination with Abraxane | Baseline up to approximately 2 years
  To measure the time from cycle 1 day 1 dose administration to the time of documented disease progression or death from any cause.
To quantify the difference in the progression free survival (PFS) in relapsed refractory metastatic breast cancer showing potentially response-predictive aberrations of MYC and other genes under ORIN1001 alone or in combination with Abraxane. | Baseline up to approximately 2 years
  To measure the time from cycle 1 day 1 dose administration to the time of documented disease progression or death from any cause.
To measure the duration of overall survival (OS) under treatment with ORIN1001 alone and in combination with Abraxane. | Baseline up to approximately 2 years
  To measure the duration of overall survival (OS) which is the time from Cycle 1 day 1 until death from any cause.
To quantify the difference in overall survival (OS) in relapsed refractory metastatic breast cancer showing potentially response-predictive aberrations of MYC and other genes under ORIN1001 alone or in combination with Abraxane | Baseline up to approximately 2 years
  To measure the duration of Overall Survival (OS) which is the time from Cycle 1 day 1 until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar F Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (20):
- United States (20):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCLA Health Burbank Specialty Care, Burbank, California
  - UCLA Health Laguna Hills Cancer Care, Laguna Hills, California
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Los Angeles (UCLA) - Jonsson Comprehensive Cancer Center (JCCC) - Oncology Center - Westwood, Westwood, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Denver, Colorado
  - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - University of Colorado Lone Tree Medical Center, Lone Tree, Colorado
  - University of Miami Hospital and Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - St Lukes Cancer Institute, Kansas City, Missouri
  - Roswell Park Comprehensive Cancer Center (RPCCC) (Roswell Park Cancer Institute (RPCI)), Buffalo, New York
  - Northwell Health, New Hyde Park, New York
  - Northwell Heath Cancer Institute, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor College of Medicine Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No